## Ahmanson/UCLA Adult Congenital Heart Disease Center

Dedicated to the Future of Children

## David Geffen School of Medicine Departments of Medicine, Pediatrics & Surgery

UCLA Centerfor the Health Sciences 650 Charles E. Young Drive South Room Å2-237CHS, Los Angeles, 90095-1679

Patient Related (310) 794-9629 \*Administrative Office (310) 825-2019 \*Far: (310) 825-6346

E-mail: ACHDC@nzednet.ucla.edu

Website: www.heart.ucla.edu/achdc

Evelyn Garcia

Date: 1 1/14/2022

Date: 1/11/2017

Sincerely,

for

Medical and Surgical Faculty

Jamil Aboulhosn, M.D., Director

Leigh Reardon, MD.

Jeannette Lin, M.D. Jeremy Moore, MD. Kevin Shannon, M.D.

Gentian Liuri, M.D., PhD Kalyanam Shivkumar, MD., PhD

Daniel Levi, M.D.

John Moriarty, M.D.

Paul Finn, M.D.

RE: A Randomized Trial of Closed Loop Stimulation after Pacemaker Implantation Pierangelo Renella, M.D.

Hillel Laks, M.D.

Brian Reemtsen, M.D.

Congenital heart Disease Reshma Biniwale, M.D. NCT: NCT03361 189 Richard Shemin, M.D. Protocol ID: 17-000932 John S. Child, M.D., Emeritus

Director

Nursing Pamela D. Miner, RN, MN, NP Linda Houser, RN, MS, NP

Jennifer Doliner, RN, BSN

Mary Canobbio, RN, MN

Social Work

David Highfill, MSW,

**LCSW** 

Research Coordinators Abbie Hageman, B.S.

Rachel Bolanos, MPH Jana

Tarabay, M.D.

Administrative Sta Yvonne Jose

Veronica Olmedo

Administrative Manager

Program

100 Medical Plaza Drive, Suite 770

Los Angeles, CA 90095

Jeremy P. Moore, MD, MS, CCDS, CEPS, FHRS

Please find attached Consents from 7/23/2018 to 3/10/2021.

Fellowship Program Director I Director of Clinical Research I Division of Pediatric Cardiology

Clinical Faculty I Ahmanson-UCLA, Adult Congenital Heart Disease

# UNIVERSITY OF CALIFORNIA LOS ANGELES CONSENT TO PARTICIPATE IN RESEARCH

A Randomized Trial of Closed Loop Stimulation after Epicardial Pacemaker Implantation for Congenital Heart Disease

#### INTRODUCTION

Jeremy P. Moore, MD MS, and associates from the Pediatric and Adult Congenital Heart Disease Program at the University of California, Los Angeles are conducting a research study.

The researchers will explain this study to you. Research studies are voluntary and include only people who choose to take part. Please take your time about deciding whether to participate in this study. Before deciding:

- You can discuss this study with friends and family.
- You can also discuss it with your health care doctor or request a second opinion. If you have any questions, you can ask the researchers for more information before deciding to participate.

The research team is asking you to be in this study because you have been identified as having congenital heart disease with a surgical pacemaker for sinus node dysfunction.

#### WHY IS THIS STUDY BEING DONE?

The purpose of this research study is to determine if a new type of pacing is helpful in terms of quality of life and exercise tolerance after cardiac surgery.

Your pacemaker company (Biotronik Inc.) has included the software for the unique pacing algorithm in all of its cardiac implantable electronic devices (i.e. pacemakers and defibrillators). The pacing algorithm is approved by the FDA, but has not been studied specifically in patients with various forms of congenital heart disease. This study is sponsored financially by Biotronik Inc.

#### WHAT WILL HAPPEN IF I TAKE PART IN THIS STUDY?

## Before you begin the study:

Before you begin the study, you will need to review this consent form carefully and decide if you are willing to participate. If you decide to participate in the study, you must sign your name and return this form to the study investigators.

## During the study:

#### D:IRB#17-000932

If you take part in this study, you will be randomly assigned to one of two possible pacemaker modes. The first pacing mode is your current pacing mode, which is based on a type of motion sensor (also known as an "accelerometer") to determine your target heart rate. The second pacing mode ("closed loop stimulation" or "CLS") relies on the pacemaker's determination of the force of contraction of your heart to estimate your target heart rate. Both pacemaker modes are FDA approved for regulation of heart rate. The second pacing mode, or "CLS" has not been studied in patients with congenital heart disease however.

At the end of 3 months, the researchers will ask you to complete a questionnaire describing your quality of life as well as perform a series of cardiac tests that include activities while wearing a gas exchange mouthpiece, testing of your autonomic nervous system function, and a mental stress test. Autonomic function testing involves testing of the unconscious part of your nervous system that is responsible for automatic activities such as regulation of heart rate, respiratory rate, digestion, and sweating, etc. This testing involves measures of blood pressure, heart rate, and sweating response to activities such as standing, deep breathing, forced exhalation (also known as a "Valsalva maneuver"). The mental stress involves completion of moderately complex mathematic problems, in order to assess your heart rate response during this type of challenge.

The time required for these activities is generally 10 minutes or less for the quality of life questionnaire, 20 minutes for exercise testing, and 30 minutes for the combination of autonomic function testing and mental stress testing (the total testing time is expected to last approximately 1 hour).

You will then be placed in the alternate pacing mode for an additional 3 months, after which all of the tests will be repeated. At the conclusion of the study, the pacing mode that is most helpful for you will be revealed, and your pacemaker will be programmed to that particular pacing mode.

#### HOW LONG WILL BE IN THIS STUDY?

This study will last 6 months.

#### WHAT KINDS OF RISKS OR DISCOMFORTS COULD I EXPECT?

#### Known risks and discomforts:

The possible risks and/or discomforts associated with the procedures described in this consent form include:

There are risks associated with exercise in patients with congenital heart disease, including the risk of provoking ventricular arrhythmia. Nevertheless, exercise testing (including gas exchange monitoring) is routinely performed as a part of the routine evaluation process and will not differ from standard testing in this study.

There is a risk of inappropriately fast pacing associated with the CLS algorithm. The degree of excessively fast pacing is limited by the study investigator at the time of pacemaker reprogramming however, so that should this occur, symptoms are expected to be limited to the sensation of palpitations. The pacemaker will not be permitted to pace your heart at dangerously fast levels on the basis of this programming.

#### Unknown risks and discomforts:

The experimental treatments may have side effects that no one knows about yet. The researchers will let you know if they learn anything that might make you change your mind about participating in the study.

#### ARE THERE ANY BENEFITS IF I PARTICIPATE?

#### Possible benefits to me:

The possible benefits you may experience from being in this study include a greater understanding of how your heart responds to different pacemaker modes. This information may be useful for future management of your cardiac pacemaker.

#### Possible benefits to others or society:

This study will help the researchers learn more about cardiac pacemakers after surgery for congenital heart disease. Hopefully this information will help in the treatment of future patients with sinus node dysfunction like yours.

#### HOW MANY PEOPLE WILL TAKE PART IN THIS STUDY?

This study will involve approximately 12 patients over the course of 5 years. Atl of the participants will have similar forms of congenital heart disease and requirements for pacemaker placement.

# WHAT OTHER CHOICES DO I HAVE IF I DON'T WANT TO PARTICIPATE?

If you decide not to take part in this study, or if you withdraw from this study before it is completed, you will continue with your current pacemaker programming and future changes will only be made as deemed necessary by your cardiac care provider.

#### CAN THE RESEARCHERS REMOVE ME FROM THIS STUDY?

The researchers may end your participation in this study for a number of reasons, such as if your safety and welfare are at risk, if you do not follow instructions or if you miss scheduled visits. The researchers or the study sponsor might also decide to stop the study at any time.

# HOW WILL INFORMATION ABOUT ME AND MY PARTICIPATION BE KEPT CONFIDENTIAL?

The researchers will do their best to make sure that your private information is kept confidential. Information about you will be handled as confidentially as possible, but participating in research may involve a loss of privacy and the potential for a breach in confidentiality. Study data will be physically and electronically secured. As with any use of electronic means to store data, there is a risk of breach of data security.

Use of personal information that can identify you:

The data used for this study will be coded so that there are no personal identifiable features directly contained within it. A code with your name will be stored separately, so that the research team can access your medical record during the study period if necessary.

How information about you will be stored:

Study data will be stored on a password encrypted research related computer server. Only the research team will have access to the data.

People and agencies that will have access to your information:

Only the research team and authorized UCLA personnel may have access to study data and records to monitor the study, Research records provided to authorized, non-UCLA personnel will not contain identifiable information about you. Publications and/or presentations that result from this study will not identify you by name.

How long information from the study will be kept:

The study data will be stored for a total of 8 years.

#### ARE THERE ANY COSTS FOR TAKING PART IN THIS STUDY?

The study will pay for the cost of all cardiac testing during the study period, and all required study items and services as described in this consent form.

#### WILL I BE PAID FOR MY PARTICIPATION?

You will not be paid for your participation in this research study.

# WHO CAN I CONTACT IF I HAVE QUESTIONS ABOUT THIS STUDY? The Research Team:

You may contact Jeremy P Moore, MD MS at 310-267-7600 with any questions or concerns about the research or your participation in this study. You can also call the UCLA Page Operator at (310) 825-6301 to reach Jeremy P. Moore or one of the covering fellows 24 hours a day, 7 days week.

## UCLA Office of the Human Research Protection Program (OHRPP):

If you have questions about your rights while taking part in this study, or you have concerns or suggestions and you want to talk to someone other than the researchers about the study, you may contact the UCLA OHRPP by phone: (310) 825-5344; by email: <a href="mailto:mirb@research.ucla.edu">mirb@research.ucla.edu</a> or U.S. mail: UCLA OHRPP, 1 1000 Kinross Ave., Suite 21 1, Box 951694, Los Angeles, CA 90095-1694.

#### Public Information about this Study:

ClinicalTrials.gov is a website that provides information about federally and privately supported clinical trials. A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

# WHAT HAPPENS IF I BELIEVE I AM INJURED BECAUSE I TOOK PART IN THIS STUDY?

It is important that you promptly tell the researchers if you believe that you have been injured because of taking part in this study. You can tell the researcher in person or call him/her at the number listed above.

If you are injured as a result of being in this study, UCLA will provide necessary medical treatment. The costs of the treatment may be covered by the University of California or the study sponsor Biotronik, or billed to you or your insurer just like other medical costs, depending on a number of factors. The University and the study sponsor do not normally provide any other form of compensation for injury. For more information about this, you may call the UCLA Office of the Human Research Protection Program at 310825-5344 or send an email to mirb@research.ucla.edu.

#### WHAT ARE MY RIGHTS IF I TAKE PART IN THIS STUDY?

Taking part in this study is your choice. You can choose whether or not you want to participate. Whatever decision you make, there wilt be no penalty to you and you will not lose any of your regular benefits.

- You have a right to have all of your questions answered before deciding whether to take part.
- Your decision will not affect the medical care you receive from UCLA.
- If you decide to take part, you can leave the study at anytime.
- If you decide to stop being in this study you should notify the research team right away. The researchers may ask you to complete some procedures in order to protect your safety.
- If you decide not to take part, you can still get medical care from UCLA.

#### HOW DO I INDICATE MY AGREEMENT TO PARTICIPATE?

If you agree to participate in this study you should sign and date below. You have been given a copy of this consent form and the Research Participant's Bill of Rights to keep. You will be asked to sign a separate form authorizing access, use, creation, or disclosure of health information about you.

# Name of Participant Signature of Participant Date SIGNATURE OF PERSON OBTAINING CONSENT Name of Person Obtaining Consent Contact Number

Date

Signature of Person Obtaining Consent

# UNIVERSITY OF CALIFORNIA LOS ANGELES CONSENT TO PARTICIPATE IN RESEARCH

A Randomized Trial of Closed Loop Stimulation after Epicardial Pacemaker Implantation for Congenital Heart Disease

#### INTRODUCTION

Jeremy P. Moore, MD MS, and associates from the Pediatric and Adult Congenital Heart Disease Program at the University of California, Los Angeles are conducting a research study.

The researchers will explain this study to you. Research studies are voluntary and include only people who choose to take part. Please take your time about deciding whether to participate in this study. Before deciding:

- You can discuss this study with friends and family.
- You can also discuss it with your health care doctor or request a second opinion.
  - If you have any questions, you can ask the researchers for more information before deciding to participate.

The research team is asking you to be in this study because you have been identified as having congenital heart disease with a surgical pacemaker for sinus node dysfunction.

#### WHY IS THIS STUDY BEING DONE?

The purpose of this research study is to determine if a new type of pacing is helpful in terms of quality of life and exercise tolerance after cardiac surgery.

Your pacemaker company (Biotronik Inc.) has included the software for the unique pacing algorithm in all of its cardiac implantable electronic devices (i.e. pacemakers and defibrillators). The pacing algorithm is approved by the FDA, but has not been studied specifically in patients with various forms of congenital heart disease. This study is sponsored financially by Biotronik Inc.

#### WHAT WILL HAPPEN IF I TAKE PART IN THIS STUDY?

## Before you begin the study:

Before you begin the study, you will need to review this consent form carefully and decide if you are willing to participate. If you decide to participate in the study, you must sign your name and return this form to the study investigators.

## During the study:

If you take part in this study, you will be randomly assigned to one of two possible pacemaker modes. The first pacing mode is your current pacing mode, which is based on a type of motion sensor (also known as an "accelerometer") to determine your target heart rate. The second pacing mode ("closed loop stimulation" or "CLS") relies on the pacemaker's determination of the force of contraction of your heart to estimate your target heart rate. Both pacemaker modes are FDA approved for regulation of heart rate. The second pacing mode, or "CLS" has not been studied in patients with congenital heart disease however.

At the end of 3 months, the researchers will ask you to complete a questionnaire describing your quality of life as well as perform a series of cardiac tests that include activities while wearing a gas exchange mouthpiece, testing of your autonomic nervous system function, and a mental stress test. Autonomic function testing involves testing of the unconscious part of your nervous system that is responsible for automatic activities such as regulation of heart rate, respiratory rate, digestion, and sweating, etc. This testing involves measures of blood pressure, heart rate, and sweating response to activities such as standing, deep breathing, forced exhalation (also known as a "Valsalva maneuver"). The mental stress involves completion of moderately complex mathematic problems, in order to assess your heart rate response during this type of challenge.

The time required for these activities is generally 10 minutes or less for the quality of life questionnaire, 20 minutes for exercise testing, and 30 minutes for the combination of autonomic function testing and mental stress testing (the total testing time is expected to last approximately 1 hour).

You will then be placed in the alternate pacing mode for an additional 3 months, after which all of the tests will be repeated. At the conclusion of the study, the pacing mode that is most helpful for you will be revealed, and your pacemaker will be programmed to that particular pacing mode.

#### HOW LONG WILL I BE IN THIS STUDY?

This study will last 6 months.

#### WHAT KINDS OF RISKS OR DISCOMFORTS COULD I EXPECT?

#### Known risks and discomforts:

The possible risks and/or discomforts associated with the procedures described in this consent form include:

There are risks associated with exercise in patients with congenital heart disease, including the risk of provoking ventricular arrhythmia. Nevertheless, exercise testing (including gas exchange monitoring) is routinely performed as a part of the routine evaluation process and will not differ from standard testing in this study.

There is a risk of inappropriately fast pacing associated with the CLS algorithm. The degree of excessively fast pacing is limited by the study investigator at the time of pacemaker reprogramming however, so that should this occur, symptoms are expected to be limited to the sensation of palpitations. The pacemaker will not be permitted to pace your heart at dangerously fast levels on the basis of this programming.

#### Unknown risks and discomforts:

The experimental treatments may have side effects that no one knows about yet. The researchers will let you know if they learn anything that might make you change your mind about participating in the study.

#### ARE THERE ANY BENEFITS IF I PARTICIPATE?

#### Possible benefits to me:

The possible benefits you may experience from being in this study include a greater understanding of how your heart responds to different pacemaker modes. This information may be useful for future management of your cardiac pacemaker.

#### Possible benefits to others or society:

This study will help the researchers learn more about cardiac pacemakers after surgery for congenital heart disease. Hopefully this information will help in the treatment of future patients with sinus node dysfunction like yours.

#### HOW MANY PEOPLE WILL TAKE PART IN THIS STUDY?

This study will involve approximately 12 patients over the course of 5 years. All of the participants will have similar forms of congenital heart disease and requirements for pacemaker placement.

# WHAT OTHER CHOICES DO I HAVE IF I DON'T WANT TO PARTICIPATE?

If you decide not to take part in this study, or if you withdraw from this study before it is completed, you will continue with your current pacemaker programming and future changes will only be made as deemed necessary by your cardiac care provider.

#### CAN THE RESEARCHERS REMOVE ME FROM THIS STUDY?

The researchers may end your participation in this study for a number of reasons, such as if your safety and welfare are at risk, if you do not follow instructions or if you miss scheduled visits. The researchers or the study sponsor might also decide to stop the study at any time.

# HOW WILL INFORMATION ABOUT ME AND MY PARTICIPATION BE KEPT CONFIDENTIAL?

The researchers will do their best to make sure that your private information is kept confidential. Information about you will be handled as confidentially as possible, but participating in research may involve a loss of privacy and the potential for a breach in confidentiality. Study data will be physically and electronically secured. As with any use of electronic means to store data, there is a risk of breach of data security.

Use of personal information that can identify you:

The data used for this study will be coded so that there are no personal identifiable features directly contained within it. A code with your name will be stored separately, so that the research team can access your medical record during the study period if necessary.

How information about you will be stored:

Study data will be stored on a password encrypted research related computer server. Only the research team will have access to the data.

People and agencies that will have access to your information:

Only the research team and authorized UCLA personnel may have access to study data and records to monitor the study. Research records provided to authorized, non-UCLA personnel will not contain identifiable information about you. Publications and/or presentations that result from this study will not identify you by name.

How long information from the study will be kept:

The study data will be stored for a total of 8 years.

#### ARE THERE ANY COSTS FOR TAKING PART 'N THIS STUDY?

The study will pay for the cost of all cardiac testing during the study period, and all required study items and services as described in this consent form.

#### WILL I BE PAID FOR MY PARTICIPATION?

You will not be paid for your participation in this research study.

# WHO CAN I CONTACT IF I HAVE QUESTIONS ABOUT THIS STUDY?

The Research Team:

You may contact Jeremy P Moore, MD MS at 310-267-7600 with any questions or concerns about the research or your participation in this study. You can also call

the UCLA Page Operator at (310) 825-6301 to reach Jeremy P. Moore or one of the covering fellows 24 hours a day, 7 days week.

## UCLA Office of the Human Research Protection Program (OHRPP):

If you have questions about your rights while taking part in this study, or you have concerns or suggestions and you want to talk to someone other than the researchers about the study, you may contact the UCLA OHRPP by phone: (310) 825-5344; by email: <a href="mailto:mirb@research.ucla.edu">mirb@research.ucla.edu</a> or U.S. mail: UCLA OHRPP, 1 1000 Kinross Ave., Suite 21 1, Box 951694, Los Angeles, CA 90095-1694.

#### Public Information about this Study:

ClinicalTrials.gov is a website that provides information about federally and privately supported clinical trials. A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

# WHAT HAPPENS IF I BELIEVE I AM INJURED BECAUSE I TOOK PART IN THIS STUDY?

It is important that you promptly tell the researchers if you believe that you have been injured because of taking part in this study. You can tell the researcher in person or call him/her at the number listed above.

If you are injured as a result of being in this study, UCLA will provide necessary medical treatment. The costs of the treatment may be covered by the University of California or the study sponsor Biotronik, or billed to you or your insurer just like other medical costs, depending on a number of factors. The University and the study sponsor do not normally provide any other form of compensation for injury. For more information about this, you may call the UCLA Office of the Human Research Protection Program at 310825-5344 or send an email to mirb@research.ucla.edu.

#### WHAT ARE MY RIGHTS IF I TAKE PART IN THIS STUDY?

Taking part in this study is your choice. You can choose whether or not you want to participate. Whatever decision you make, there will be no penalty to you and you will not lose any of your regular benefits.

- You have a right to have all of your questions answered before deciding whether to take part.
- Your decision will not affect the medical care you receive from UCLA.
- If you decide to take part, you can leave the study at anytime.
- If you decide to stop being in this study you should notify the research team right away. The researchers may ask you to complete some procedures in order to protect your safety.

• If you decide not to take part, you can still get medical care from UCLA.

## HOW DO I INDICATE MY AGREEMENT TO PARTICIPATE?

If you agree to participate in this study you should sign and date below. You have been given a copy of this consent form and the Research Participant's Bill of Rights to keep. You will be asked to sign a separate form authorizing access, use, creation, or disclosure of health information about you.

| SIGNATURE OF THE PARTICIPANT | | |
|---------------------------------------|---------|----------|
| Name of Participant | | |
| Signature of Participant | Date | <u> </u> |
| SIGNATURE OF PERSON OBTAINING | | |
| Name of Person Obtaining Consent | Contact | |
| CONSENT | Number | |
| Signature of Person Obtaining Consent | Date | |

# UNIVERSITY OF CALIFORNIA LOS ANGELES CONSENT TO PARTICIPATE IN RESEARCH

A Randomized Trial of Closed Loop Stimulation after Epicardial Pacemaker Implantation for Congenital Heart Disease

#### INTRODUCTION

Jeremy P. Moore, MD MS, and associates from the Pediatric and Adult Congenital Heart Disease Program at the University of California, Los Angeles are conducting a research study.

The researchers will explain this study to you. Research studies are voluntary and include only people who choose to take part. Please take your time about deciding whether to participate in this study. Before deciding:

- You can discuss this study with friends and family.
- You can also discuss it with your health care doctor or request a second opinion.
- If you have any questions, you can ask the researchers for more information before deciding to participate.

The research team is asking you to be in this study because you have been identified as having congenital heart disease with a surgical pacemaker for sinus node dysfunction.

#### WHY IS THIS STUDY BEING DONE?

The purpose of this research study is to determine if a new type of pacing is helpful in terms of quality of life and exercise tolerance after cardiac surgery.

Your pacemaker company (Biotronik Inc.) has included the software for the unique pacing algorithm in all of its cardiac implantable electronic devices (i.e. pacemakers and defibrillators). The pacing algorithm is approved by the FDA, but has not been studied specifically in patients with various forms of congenital heart disease. This study is sponsored financially by Biotronik Inc.

WHAT WILL HAPPEN IF I TAKE PART IN THIS STUDY? Before you begin the study:

Before you begin the study, you will need to review this consent form carefully and decide if you are willing to participate. If you decide to participate in the study, you must sign your name and return this form to the study investigators.

#### During the study:

If you take part in this study, you will be randomly assigned to one of two possible pacemaker modes. The first pacing mode is your current pacing mode, which is based on a type of motion sensor (also known as an "accelerometer") to determine your target heart rate. The second pacing mode ("closed loop stimulation" or "CLS") relies on the pacemaker's determination of the force of contraction of your heart to estimate your target heart rate. Both pacemaker modes are FDA approved for regulation of heart rate. The second pacing mode, or "CLS" has not been studied in patients with congenital heart disease however.

At the end of 3 months, the researchers will ask you to complete a questionnaire describing your quality of life as well as perform a series of cardiac tests that include activities while wearing a gas exchange mouthpiece, testing of your autonomic nervous system function, and a mental stress test. Autonomic function testing involves testing of the unconscious part of your nervous system that is responsible for automatic activities such as regulation of heart rate, respiratory rate, digestion, and sweating, etc. This testing involves measures of blood pressure, heart rate, and sweating response to activities such as standing, deep breathing, forced exhalation (also known as a "Valsalva maneuver"). The mental stress involves completion of moderately complex mathematic problems, in order to assess your heart rate response during this type of challenge.

The time required for these activities is generally 10 minutes or less for the quality of life questionnaire, 20 minutes for exercise testing, and 30 minutes for the combination of autonomic function testing and mental stress testing (the total testing time is expected to last approximately 1 hour).

You will then be placed in the alternate pacing mode for an additional 3 months, after which all of the tests will be repeated. At the conclusion of the study, the pacing mode that is most helpful for you will be revealed, and your pacemaker will be programmed to that particular pacing mode.

#### HOW LONG WILL I BE IN THIS STUDY?

This study will last 6 months.

#### WHAT KINDS OF RISKS OR DISCOMFORTS COULD I EXPECT?

#### Known risks and discomforts:

The possible risks and/or discomforts associated with the procedures described in this consent form include:

There are risks associated with exercise in patients with congenital heart disease, including the risk of provoking ventricular arrhythmia. Nevertheless, exercise testing (including gas exchange monitoring) is routinely performed as a part of the routine evaluation process and will not differ from standard testing in this study.

There is a risk of inappropriately fast pacing associated with the CLS algorithm. The degree of excessively fast pacing is limited by the study investigator at the time of pacemaker reprogramming however, so that should this occur, symptoms are expected to be limited to the sensation of palpitations. The pacemaker will not be permitted to pace your heart at dangerously fast levels on the basis of this programming.

#### Unknown risks and discomforts:

The experimental treatments may have side effects that no one knows about yet. The researchers will let you know if they learn anything that might make you change your mind about participating in the study.

#### ARE THERE ANY BENEFITS IF I PARTICIPATE?

#### Possible benefits to me:

The possible benefits you may experience from being in this study include a greater understanding of how your heart responds to different pacemaker modes. This information may be useful for future management of your cardiac pacemaker.

### Possible benefits to others or society:

This study will help the researchers learn more about cardiac pacemakers after surgery for congenital heart disease. Hopefully this information will help in the treatment of future patients with sinus node dysfunction like yours.

#### HOW MANY PEOPLE WILL TAKE PART IN THIS STUDY?

This study will involve approximately 12 patients over the course of 5 years. All of the participants will have similar forms of congenital heart disease and requirements for pacemaker placement.

# WHAT OTHER CHOICES DO I HAVE IF I DON'T WANT TO PARTICIPATE?

If you decide not to take part in this study, or if you withdraw from this study before it is completed, you will continue with your current pacemaker programming and future changes will only be made as deemed necessary by your cardiac care provider.

#### CAN THE RESEARCHERS REMOVE ME FROM THIS STUDY?

The researchers may end your participation in this study for a number of reasons, such as if your safety and welfare are at risk, if you do not follow instructions or if you miss scheduled visits. The researchers or the study sponsor might also decide to stop the study at any time.

# HOW WILL INFORMATION ABOUT ME AND MY PARTICIPATION BE KEPT CONFIDENTIAL?

The researchers will do their best to make sure that your private information is kept confidential. Information about you will be handled as confidentially as possible, but participating in research may involve a loss of privacy and the potential for a breach in confidentiality. Study data will be physically and electronically secured. As with any use of electronic means to store data, there is a risk of breach of data security.

Use of personal information that can identify you:

The data used for this study will be coded so that there are no personal identifiable features directly contained within it. A code with your name will be stored separately, so that the research team can access your medical record during the study period if necessary.

How information about you will be stored:

Study data will be stored on a password encrypted research related computer server. Only the research team will have access to the data.

People and agencies that will have access to your information:

Only the research team and authorized UCLA personnel may have access to study data and records to monitor the study. Research records provided to authorized, non-UCLA personnel will not contain identifiable information about you. Publications and/or presentations that result from this study will not identify you by name.

How long information from the study will be kept:

The study data will be stored for a total of 8 years.

#### ARE THERE ANY COSTS FOR TAKING PART IN THIS STUDY?

The study will pay for the cost of all cardiac testing during the study period, and all required study items and services as described in this consent form.

#### WILL I BE PAID FOR MY PARTICIPATION?

You will not be paid for your participation in this research study.

# WHO CAN I CONTACT IF I HAVE QUESTIONS ABOUT THIS STUDY? The Research Team:

You may contact Jeremy P Moore, MD MS at 310-267-7600 with any questions or concerns about the research or your participation in this study. You can also call the UCLA Page Operator at (310) 825-6301 to reach Jeremy P. Moore or one of the covering fellows 24 hours a day, 7 days week.

## UCLA Office of the Human Research Protection Program (OHRPP):

If you have questions about your rights while taking part in this study, or you have concerns or suggestions and you want to talk to someone other than the researchers about the study, you may contact the UCLA OHRPP by phone: (310) 825-5344; by email: <a href="mailto:mirb@research.ucla.edu">mirb@research.ucla.edu</a> or U.S. mail: UCLA OHRPP, 11000 Kinross Ave., Suite 211, Box 951694, Los Angeles, CA 90095-1694.

#### Public Information about this Study:

ClinicalTrials.gov is a website that provides information about federally and privately supported clinical trials. A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

# WHAT HAPPENS IF I BELIEVE I AM INJURED BECAUSE I TOOK PART IN THIS STUDY?

It is important that you promptly tell the researchers if you believe that you have been injured because of taking part in this study. You can tell the researcher in person or call him/her at the number listed above.

If you are injured as a result of being in this study, UCLA will provide necessary medical treatment. The costs of the treatment may be covered by the University of California or the study sponsor Biotronik, or billed to you or your insurer just like other medical costs, depending on a number of factors. The University and the study sponsor do not normally provide any other form of compensation for injury. For more information about this, you may call the UCLA Office of the Human Research Protection Program at 310825-5344 or send an email to <a href="mailto:mirb@research.ucla.edu">mirb@research.ucla.edu</a>.

#### WHAT ARE MY RIGHTS IF TAKE PART IN THIS STUDY?

Taking part in this study is your choice. You can choose whether or not you want to participate. Whatever decision you make, there will be no penalty to you and you will not lose any of your regular benefits.

- You have a right to have all of your questions answered before deciding whether to take part.
- Your decision will not affect the medical care you receive from UCLA.
- If you decide to take part, you can leave the study at anytime.
- If you decide to stop being in this study you should notify the research team right away. The researchers may ask you to complete some procedures in order to protect your safety.
- If you decide not to take part, you can still get medical care from UCLA.

## HOW DO I INDICATE MY AGREEMENT TO PARTICIPATE?

If you agree to participate in this study you should sign and date below. You have been given a copy of this consent form and the Research Participant's Bill of Rights to keep. You will be asked to sign a separate form authorizing access, use, creation, or disclosure of health information about you.

## SIGNATURE OF THE PARTICIPANT

| Name of Participant | | |
|------------------------------------------|-------------------|---|
| Signature of Participant | Date | |
| SIGNATURE OF PERSON OBTAINING<br>CONSENT | | |
| Name of Person Obtaining Consent | Contact<br>Number | |
| Signature of Person Obtaining Consent | Date | · |